CLINICAL TRIAL: NCT06202326
Title: Role of Renal Artery Doppler In Critically Ill Children With Acute Kidney Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nardeen Emad Elway, assistant lecturer, Assiut University
Other Study IDs: AKI in critically ill children
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: renal artery doppler — doppler ultrasound follow up

SUMMARY:
To detect frequency of acute kidney injury in critically ill children in Assuit university hospital.

To detect associated AKI risk factors, severity and outcomes . To assess the value of use of renal Doppler ultrasound in AKI.

DETAILED DESCRIPTION:
Critically ill child is defined as a child whose baseline state of health has significantly changed and whose life is at risk as a result of an illness or injury and they in big need for intensive care whether medicallyor surgically.

Acute kidney injury (AKI) is characterized by a sudden and generally revertible renal function impairment , involving inability to maintain the homeostasis, and may or not be accompanied by reduced diuresis. (1) Acute kidney injury (AKI) is highly prevalent among hospitalized children, with incidence rates ranging from 5% in non-critically ill children to 50% in those admitted to pediatric emergency units (2). This disease is strongly associated with worse outcomes, including increased mortality, increased use of mechanical ventilation, and prolonged hospital stay (3). AKI prevalence due to sepsis ranges from 9% to 40%, involves poor prognosis, and is associated with a 70% mortality rate (4). Among critically ill renal impaired patients, about 6% the septic shock, is one of the main causes of AKI. may need renal replacement therapy (RRT), with a mortality rate increased by 50 to 80%, particularly associated with sepsis, septic shock, and multiple organ and systems dysfunction MODS (5).

During the childhood, the main AKI causes are sepsis, nephrotoxic drugs, and renal ischemia in critically ill patients (1) .These patients, particularly those staying in intensive care units , are exposed to a number of conditions which may result in renal impairment ,thus significantly increasing the morbidity and mortality rate. (6).

Among the main causes that should be mentioned : hypovolemia leading to hypoperfusion and consequent hypoxia; inflammatory and thrombotic events caused by bacteremia ; systemic inflammation from trauma, major surgeries, extracorporeal circulation ;use of vasodilator drugs such as phosphodiesterase inhibitors, sedatives, epidural blockade; vasopressors; and use of nephrotoxic drugs as aminoglycosides, amphotericin B, radiological contrasts, and drugs interfering with the renal hemodynamics such as angiotensin converting enzyme inhibitors and angiotensin II receptor blockers (3).

In 2004, a consensus definition for AKI was proposed by the Acute Dialysis Quality Initiative (ADQI) : the RIFLE criteria (risk, injury ,failure, loss, end-stage renal disease) (7) .The adult-derived RIFLE definition was modified, and then applied and validated in pediatric patients and renamed as the pediatric RIFLE criteria. pRIFLE stratifies AKI from mild (RIFLE R, risk) to severe (RIFLE F, failure) based on changes in SCR or estimated creatinine clearance and urine output .Similar to adult studies AKI defined by these criteria was an independent risk factor for both increased hospital length of stay and mortality.

Currently, the most widely used criteria for diagnosing and staging AKI is the Kidney Disease Improving Global Outcomes (KDIGO) criteria, which is based on acute changes in serum creatinine (sCr) and/or reduced urine output (UO) (8). These criteria have limitations, especially in children. Significant sCr elevations can be delayed 24 to 48 hours after a renal insult and are commonly seen only after at least 50% of renal function loss. In addition, children may have very low sCr levels at baseline, which can make it difficult to identify relative increases when values remain within normal ranges. To overcome these limitatio, point-of-care ultrasonography has been proposed as a reliable and safe method to both diagnose and predict the occurrence of AKI in ICU patients (8).

The AKI diagnosis methods include: clinical evaluation of the urine output and laboratory tests as urine analysis, blood urea nitrogen, and creatinine, however with low sensitivity and specificity.(9). Biomarkers for early AKI detection are currently under investigation, among them neutrophil gelatinase associated lipocalin (NGAL), cystatin C, interleukin 18, and kidney injury molecule-1(KIM1). Although these markers have good sensitivity and specificity, they are not routinely used due to their low availability and high costs(10). So there is a need for a method valid ,early, simple for early detection of AKI.

Renal arterial Doppler-based parameters, such as renal resistive index (RRI) or renal pulsatility index (RPI), are rapid, noninvasive, and repeatable variables that may be promising for early AKI detection. Because it reflects resistance to blood flow, lower RRI values are associated with better renal perfusion, while increased values are associated with progression to ATN (11). However, there is a lack of evidence supporting the use of this technique in PICU. Therefore, this study aims to assess the accuracy of renal arterial Doppler ultrasound (RDU) to predict AKI in mechanically ventilated children.

The complement system, which is a part of the innate immune system, is involved in mechanism of AKI , and thus could present a unifying therapeutic target in the pathophysiology of AKI development in children who are critically ill. The complement cascade is made up of three activation pathways: classic, alternative, and lectin. These three pathways feed into the "terminal complement cascade." These pathways generate protein fragments that can be quantified to determine the level of complement activation in each pathway in a given disease: C4a (classic and lectin pathways), Factors Ba and Bb (alternative pathway), C3a (all three pathways), and sC5b-9 (terminal pathway). The kidney is particularly susceptible to complement activation because complement proteins are concentrated in the kidney via glomerular filtration and activation is promoted via the kidney's acidic environment and ammonia synthesis (12). Complement factors have been shown to be instrumental in the pathogenesis of AKI in basic science models of sepsis and ischemia reperfusion injury (13,14). All three pathways have been implicated in the pathogenesis of a wide variety of kidney diseases (11,15,16).

ELIGIBILITY:
Inclusion Criteria:

1. Critically ill children aged more than 1 month up to 18 years who were admitted in Assuit University Children Hospital.
2. Critically ill and admitted in emergency unit more than 24hrs

   -

Exclusion Criteria:

* 1- Neonates ( age less than 1months) and adults (more than 18years). 2- Patient with chronic kidney disease on dialysis. 3- Patient with hospital stay duration less 24 hrs. 4- Patient with congenital kidney disease

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: critically ill children in emergency unit and PICU.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
early detection of AKI in critically ill children | baseline
  renal artery doppler can help in detection of AKI in early stage by calculate renal resistive index and renal pulsaltility index

IPD SHARING:
Plan to Share IPD: Undecided